CLINICAL TRIAL: NCT02342886
Title: A Phase 3 Open-Label Partially Randomized Trial to Evaluate the Efficacy, Safety and Tolerability of the Combination of Moxifloxacin Plus PA-824 Plus Pyrazinamide After 4 and 6 Months of Treatment in Adult Subjects With Drug-Sensitive Smear-Positive Pulmonary Tuberculosis and After 6 Months of Treatment in Adult Subjects With Multi-Drug Resistant, Smear-Positive Pulmonary Tuberculosis.
Brief Title: Shortening Treatment by Advancing Novel Drugs
Acronym: STAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC-006-(M-PA-Z)
Record Dates: First submitted 2014-10-14; First posted 2015-01-21 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Tuberculosis, Pulmonary, Drug Sensitive; Tuberculosis, Pulmonary, Multi Drug-resistant
Keywords: Tuberculosis; Multi Drug-Resistant Tuberculosis; Drug-sensitive Tuberculosis; PA-824; Moxifloxacin; Pyrazinamide; Rifampicin; Isoniazid; Ethambutol; HRZE; HR; Pretomanid; NC-006; STAND
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — Moxifloxacin; pretomanid; Pyrazinamide; Rifampin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MDR-TB (Experimental): moxifloxacin 400 mg + PA-824 200 mg + pyrazinamide 1500 mg for 26 weeks.
  Interventions: Drug: Moxifloxacin; Drug: PA-824; Drug: Pyrazinamide
- DS-TB (HRZE), HR (Active Comparator): 26 consecutive weeks to DS-TB subjects only, as follows:
  HRZE (Rifampicin, Isoniazid, Pyrazinamide, Ethambutol combination) Weeks 1-8 with daily dose per the subjects weight
  HR (Rifampicin plus isoniazid combination tablets) Weeks 9 - 26 with daily dose per the subjects weight
  Daily dose per the subjects weight as follows: 30-39kg: 2 tablets; 40-54kg: 3 tablets; 55 - 70kg: 4 tablets; 71kg and over: 5 tablets.
  Interventions: Drug: HRZE (Rifampicin, Isoniazid, Pyrazinamide, Ethambutol combination); Drug: HR (rifampicin plus isoniazid combination tablets)
- DS-TB PA-824 200mg 26 weeks (Experimental): moxifloxacin 400 mg + PA-824 200 mg + pyrazinamide 1500 mg orally once daily for 26 weeks
  Interventions: Drug: Moxifloxacin; Drug: PA-824; Drug: Pyrazinamide
- DS-TB PA-824 200mg 17 weeks (Experimental): moxifloxacin 400 mg + PA-824 200 mg + pyrazinamide 1500 mg orally once a day for 17 weeks
  Interventions: Drug: Moxifloxacin; Drug: PA-824; Drug: Pyrazinamide
- DS-TB PA-824 100mg 17 weeks (Experimental): moxifloxacin 400 mg + PA-824 100 mg + pyrazinamide 1500 mg orally once daily for 17 weeks
  Interventions: Drug: Moxifloxacin; Drug: PA-824; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Moxifloxacin — Oral
  Other Names: BAY 12-8039; Avelox; Avalon; Avelon
  Arms: DS-TB PA-824 100mg 17 weeks; DS-TB PA-824 200mg 17 weeks; DS-TB PA-824 200mg 26 weeks; MDR-TB
Drug: PA-824 — Oral
  Arms: DS-TB PA-824 100mg 17 weeks; DS-TB PA-824 200mg 17 weeks; DS-TB PA-824 200mg 26 weeks; MDR-TB
Drug: Pyrazinamide — Oral
  Arms: DS-TB PA-824 100mg 17 weeks; DS-TB PA-824 200mg 17 weeks; DS-TB PA-824 200mg 26 weeks; MDR-TB
Drug: HRZE (Rifampicin, Isoniazid, Pyrazinamide, Ethambutol combination) — Oral
  Other Names: Rifafour e-275
  Arms: DS-TB (HRZE), HR
Drug: HR (rifampicin plus isoniazid combination tablets) — Oral
  Arms: DS-TB (HRZE), HR

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of a combination of moxifloxacin, PA-824, and pyrazinamide treatments with varying doses and treatment lengths from 4 to 6 months in subjects with drug-sensitive (DS) pulmonary TB compared to standard HRZE treatment.

This study will also assess the efficacy, safety and tolerability of a combination of moxifloxacin, PA-824, and pyrazinamide treatments after 6 months of treatment in subjects with multi drug-resistant (MDR) pulmonary TB compared to a combination of moxifloxacin, PA-824, and pyrazinamide treatments in DS-TB subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written consent or witnessed oral consent in the case of illiteracy, prior to undertaking any trial-related procedures.
2. Male or female, aged 18 years or over.
3. Body weight (in light clothing and no shoes) ≥ 30 kg.
4. Sputum positive for tubercule bacilli (at least 1+ on the International Union Against Tuberculosis and Lung Disease (IUATLD) and World Health Organization (WHO) scale on smear microscopy at the trial laboratory.
5. Drug-Sensitive TB treatment arms subjects should be:

   * sensitive to rifampicin by rapid sputum based test (may be sensitive or resistant to isoniazid) AND
   * either newly diagnosed for TB or have a patient history of being untreated for at least 3 years after cure from a previous episode of TB. If they are entered into the trial due to being sensitive to rifampicin by rapid sputum based test, however on receipt of the rifampicin resistance testing using an indirect susceptibility test in liquid culture this shows they are rifampicin resistant, they will be:
   * Excluded as late exclusions;
   * Possibly replaced as determined by the sponsor.
6. MDR-TB treatment arm subjects should be resistant to rifampicin by rapid sputum based test (may be sensitive or resistant to isoniazid).
7. A chest x-ray which in the opinion of the investigator is compatible with pulmonary TB.
8. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

* Subject - not heterosexually active or practice sexual abstinence; or
* Female subject or male subjects female sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months; or
* Male subject or female subjects male sexual partner - vasectomised or has had a bilateral orchidectomy minimally three months prior to screening;

Effective birth control methods:

* Double barrier method which can include a male condom, diaphragm, cervical cap, or female condom; or
* Female subject: Barrier method combined with hormone-based contraceptives or an intra-uterine device for the female patient.
* Male subjects' female sexual partner: Double barrier method or hormone-based contraceptives or an intra-uterine device for the female partner.

and are willing to continue practising birth control methods and are not planning to conceive throughout treatment and for 12 weeks (male subjects) or 1 week (female subjects) after the last dose of trial medication or discontinuation from trial medication in case of premature discontinuation.

(Note: Hormone-based contraception alone may not be reliable when taking IMP; therefore,

Exclusion Criteria:

1. Any non TB related condition (including myasthenia gravis) where participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments.
2. Being or about to be treated for Malaria.
3. Is critically ill and, in the judgment of the investigator, has a diagnosis likely to result in death during the trial or the follow-up period.
4. TB meningitis or other forms of extrapulmonary tuberculosis with high risk of a poor outcome, or likely to require a longer course of therapy (such as TB of the bone or joint), as judged by the investigator.
5. History of allergy or hypersensitivity to any of the trial IMP or related substances, including known allergy to any fluoroquinolone antibiotic, history of tendinopathy associated with quinolones or suspected hypersensitivity to any rifampicin antibiotics.
6. For HIV infected subjects any of the following:

   * CD4+ count <100 cells/µL;
   * Karnofsky score <60%;
   * Received intravenous antifungal medication within the last 90 days;
   * WHO Clinical Stage 4 HIV disease.
7. Resistant to fluoroquinolones (rapid, sputum - based molecular screening tests). If they are entered into the trial due to being sensitive to fluoroquinolones by rapid sputum based test, however on receipt of the fluoroquinolones resistance testing using an indirect susceptibility test in liquid culture this shows they are fluoroquinolones resistant, they will be:

   * Excluded as late exclusions;
   * Possibly replaced as determined by the sponsor.
8. Resistant to pyrazinamide (rapid, sputum - based molecular screening tests).

   Drug-Sensitive TB treatment arms subjects may be entered prior to receipt of the rapid, sputum - based molecular pyrazinamide resistance screening test result. On receipt of the result, if they are resistant, they will be:
   * Excluded as late exclusions;
   * Possibly replaced as determined by the sponsor. MDR-TB treatment arm subjects may not be entered prior to receipt of the rapid, sputum - based molecular pyrazinamide resistance screening test result showing they are sensitive to pyrazinamide.
9. Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
10. Subjects with any of the following at screening (per measurements and reading done by Central Electrocardiogram (ECG) where applicable):

    * Cardiac arrhythmia requiring medication;
    * Prolongation of QT/QTc interval with QTcF (Fridericia correction) >450 ms;
    * History of additional risk factors for Torsade de Pointes, (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
    * Any clinically significant ECG abnormality, in the opinion of the investigator.
11. Unstable Diabetes Mellitus which required hospitalization for hyper- or hypo-glycaemia within the past year prior to start of screening.

    Specific Treatments
12. Previous treatment with PA-824 as part of a clinical trial.
13. For DS-TB treatment arms: Previous treatment for tuberculosis within 3 years prior to Day (-9 to -1)(Screening). Subjects who have previously received isoniazid prophylactically may be included in the trial as long as that treatment is/was discontinued at least 7 days prior to randomization into this trial.

    For the MDR-TB Subjects: Previous treatment for MDR-TB, although may have been on a MDR TB treatment regimen for no longer than 7 days at start of screening.

    Previous treatment for TB includes, but is not limited to, gatifloxacin, amikacin, cycloserine, rifabutin, kanamycin, para-aminosalicylic acid, rifapentine, thioacetazone, capreomycin, quinolones, thioamides, and metronidazole.
14. Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.
15. Use of any drug within 30 days prior to randomisation known to prolong QTc interval (including, but not limited to, amiodarone, amitriptyline, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinacrine, quinidine, sotalol, sparfloxacin, thioridazine).
16. Use of systemic glucocorticoids within one year of start of screening (inhaled or intranasal glucocorticoids are allowed).
17. Subjects recently started or expected to need to start anti-retroviral therapy (ART) within 1 month after randomization. Subjects may be included who have been on ARTs for greater than 30 days prior to start of screening, or who are expected to start ART greater than 30 days after randomization.

    Laboratory Abnormalities
18. Subjects with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007), where applicable:

    * creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    * creatinine clearance (CrCl) level less than 30 mLs/min according to the Cockcroft-Gault Formula;
    * haemoglobin grade 4 (<6.5 g/dL);
    * platelets grade 3 or greater (under 50x109 cells/L/ 50 000/mm3);
    * serum potassium less than the lower limit of normal for the laboratory. This may be repeated once;
    * aspartate aminotransferase (AST) grade 3 or greater (≥3.0 x ULN) ;
    * alanine aminotransferase (ALT) grade 3 or greater (≥3.0 x ULN);
    * alkaline phosphatase (ALP):

      * grade 4 (>8.0 x ULN) to be excluded;
      * grade 3 (≥3.0 - 8.0 x ULN) must be discussed with and approved by the sponsor Medical Monitor;
    * total bilirubin:

      * 2.0 x ULN, when other liver functions are in the normal range
      * 1.50 x ULN when accompanied by any increase in other liver function tests subjects with total bilirubin > 1.25 x ULN and accompanied by any increase in other liver function tests must be discussed with the sponsor medical monitor before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Gillespie, MD, Principal Investigator — University of St Andrews
Locations (26):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Kenya (2):
  - Centre for Respiratory Disease Research (CRDR) Keny Medical Research Institute (KEMRI), Nairobi
  - Centre for Respiratory Disease Research (CRDR) Kenya Medical Research Institute (KEMRI), Nairobi
- Malaysia (3):
  - Pusat Perubatan Universiti Kebangsaan, Cheras, Kuala Lumpur
  - Universiti Teknologi MARA, Batu Caves, Selangor
  - Institute of Respiratory Medicine (IPR), Kuala Lumpur
- Philippines (3):
  - Philippine General Hospital, Ermita, Manila
  - Vincent Balang, Pio del Pilar, Manila
  - Lung Center of Philippines, Manila
- South Africa (12):
  - TASK, Bellville, Cape Town
  - University of Cape Town Lung Institute, Mowbray, Cape Town
  - Setshaba Research Centre, Pretoria, Gauteng
  - The Aurum Institute: Tembisa Hospital Cnr, Tembisa, Gauteng
  - CHRU Themba Lethu Clinic, Westdene, Johannesburg
  - Durban International Clinical Trials Unit (DbnlCTU), Durban, KwaZulu-Natal
  - Klerksdorp Tshepong Hospital, Klerksdorp, North West
  - Synexus SA, Mamelodi East, Pretoria
  - Madibeng Centre for Research (MCR), Brits
  - THINK: Tuberculosis & HIV Investigative Network of Kwazulu Natal, Durban
  - The Aurum Institute, Klerksdorp
  - The Aurum Institute: Rustenberg, Rustenburg
- Tanzania (3):
  - Ifakara Health Institute (IHI), Dar es Salaam
  - NIMR - Mbeya Medical Research Programme (MMRP), Mbeya
  - Kilimanjaro National Institute for Medical Research, Mwanza
- Uganda CWRU Research Collaboration, Kampala, Uganda
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female patients with drug-sensitive (DS) and multi-drug resistant (MDR) smear-positive pulmonary tuberculosis (TB) were recruited into this open-label multicenter study.
Pre-assignment Details: Patients were confirmed sputum positive for tubercule bacilli on smear microscopy. DS-TB patients were required to be sensitive to rifampicin and newly diagnosed with pulmonary TB (or untreated for at least 3 years). MDR-TB patients were required to be resistant to rifampicin. Both DS and MDR-TB patients could be sensitive/resistant to isoniazid.
Groups:
- DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide: Patients with DS-TB were randomized to receive 400 milligrams (mg) moxifloxacin + 100 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 4 months during the treatment period (from Day 1 to Week 17). Patients then entered a follow-up period up to Month 24.
- DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide: Patients with DS-TB were randomized to receive 400 mg moxifloxacin + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 4 months during the treatment period (from Day 1 to Week 17). Patients then entered a follow-up period up to Month 24.
- DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide: Patients with DS-TB were randomized to receive 400 mg moxifloxacin + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 6 months during the treatment period (from Day 1 to Week 26). Patients then entered a follow-up period up to Month 24.
- DS-TB: 2 Months HRZE / 4 Months HR: Patients with DS-TB were randomized to receive 150 mg rifampicin + 75 mg isoniazid + 400 mg pyrazinamide + 275 mg ethambutol combination tablets (HRZE) orally once daily from Weeks 1 to 8 during the treatment period. Patients then received 150 mg rifiampicin + 75 mg isoniazid combination tablets (HR) orally once daily from Weeks 9 to 26 during the treatment period. The daily dose of HRZE and HR was calculated based on patients' weight. Patients then entered a follow-up period up to Month 24.
- MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide: Patients with MDR-TB received 400 mg moxifloxacin + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 6 months during the treatment period (from Day 1 to Week 26). Patients then entered a follow-up period up to Month 24.
Period: Overall Study
Arm/Group | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 2 Months HRZE / 4 Months HR | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide
Started | 65 | 71 | 67 | 68 | 13
Completed Month 12 Follow-Up | 43 | 52 | 49 | 57 | 10
Completed Month 24 Follow-Up | 40 | 47 | 46 | 53 | 10
Completed (Completed Treatment) | 57 | 63 | 52 | 59 | 10
Not Completed | 8 | 8 | 15 | 9 | 3
Not completed — Treatment non-compliance | 1 | 0 | 0 | 1 | 0
Not completed — Late exclusion: rifampicin resistance | 1 | 0 | 0 | 0 | 0
Not completed — Adverse event/specific toxicity | 4 | 3 | 11 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0
Not completed — Investigator/sponsor decision | 0 | 2 | 0 | 3 | 1
Not completed — Pregnancy | 0 | 0 | 2 | 0 | 0
Not completed — Late exclusion: pyrazinamide resistance | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis population included all patients who were randomized (for the DS-TB patients) or assigned (for the MDR-TB patients) to trial medication and who received at least 1 dose of trial medication. Patients were classified according to treatment received.
Groups:
- DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide: Patients with DS-TB were randomized to receive 400 mg moxifloxacin + 100 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 4 months during the treatment period (from Day 1 to Week 17). Patients then entered a follow-up period up to Month 24.
- Total: Total of all reporting groups
Arm/Group | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 2 Months HRZE / 4 Months HR | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | Total
Number analyzed (Participants) | 65 | 71 | 67 | 68 | 13 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 2 | 0 | 0 | 6
  Between 18 and 65 years | 63 | 67 | 65 | 67 | 13 | 275
  >=65 years | 0 | 2 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 23 | 20 | 7 | 87
  Male | 51 | 48 | 44 | 48 | 6 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 65 | 71 | 67 | 68 | 13 | 284
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 6 | 6 | 4 | 0 | 19
  Black or African American | 45 | 49 | 45 | 44 | 8 | 191
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 3 | 3 | 2 | 14
  Mixed Race | 8 | 12 | 8 | 13 | 3 | 44
  Other | 6 | 1 | 5 | 3 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Combined Bacteriologic Failure or Relapse or Clinical Failure at Month 12 From Start of Therapy (Day 1) (Modified Intent to Treat [MITT] Population)
Description: Patients were classified as having a favorable, unfavorable or unassessable status at 12 months from the start of therapy.
  A favourable status was a negative culture status at 12 months from start of therapy in patients who had not already been classified as having an unfavorable outcome, and whose last positive culture result was followed by at least 2 negative culture results. Patients with an unfavorable status did not achieve/maintain culture negative status, or previously had culture negative status who following end of treatment (EOT), had 2 positive cultures, or had a positive culture not followed by 2 negative cultures, or were dying from any cause during treatment (except accidental cause not including suicide), or were dying from TB related causes during follow-up, or required an extension, restart or change of treatment except for reinfection/pregnancy, or failed to complete adequate treatment who were unassessable at 12 months or lost to follow-up/withdrawn before EOT.
Time Frame: From Day 1 to Month 12.
Population: The MITT population included all randomized patients excluding late screening failures, lost to follow-up/withdrawn patients who were culture negative, pregnancy, accidental death during treatment, death during follow-up without TB relapse evidence, re-infection with new TB strain + missing/contaminated Month 12 sputum sample.
Measure: Count of Participants; unit: Participants
Groups:
- MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide: Patients with MDR-TB received 400 mg moxifloxacin + 200 mg pretomanid (PA-824) + 1500 mg pyrazinamide orally once daily for 6 months during the treatment period (from Day 1 to Week 26). Patients then entered a follow-up period up to Month 24.
  Note: The MDR-TB group was not randomized and not included in the analysis population.
Arm/Group | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 2 Months HRZE / 4 Months HR | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide
Number analyzed (Participants) | 57 | 61 | 56 | 60 | 11
Participants
  Favorable | 38 | 46 | 43 | 52 | 10
  Unfavorable | 19 | 15 | 13 | 8 | 1
Statistical Analysis 1: Comparison: DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide vs DS-TB: 2 Months HRZE / 4 Months HR; Test type: Non-Inferiority — Non-inferiority was assessed using the upper bound of the two-sided 95% confidence interval (CI) for the difference between the percentage of patients who are classified as having an unfavourable status on the intervention (6 months moxifloxacin + 200 mg PA-824 + pyrazinamide) and the control regimen (2 months HRZE/ 4 months HR). The intervention was considered to be non-inferior to the control arm if the upper bound 95% CI was < 12%; Treatment difference: unfavourable rate = 9.88, 95% CI 2-sided [-4.13 to 23.89] — (DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide) - (DS-TB: 2 Months HRZE/ 4 Months HR)

2. Primary Outcome: Incidence of Combined Bacteriologic Failure or Relapse or Clinical Failure at Month 12 From Start of Therapy (Day 1) (Per Protocol [PP] Population)
Description: Patients were classified as having a favorable, unfavorable or unassessable status at 12 months from the start of therapy.
  A favourable status was a negative culture status at 12 months from start of therapy in patients who had not already been classified as having an unfavorable outcome, and whose last positive culture result was followed by at least 2 negative culture results. Patients with an unfavorable status did not achieve/maintain culture negative status, or previously had culture negative status who following EOT, had 2 positive cultures, or had a positive culture not followed by 2 negative cultures, or died from any cause during treatment (except accidental cause not including suicide), or were dying from TB related causes during follow-up, or required a restart or change of treatment because of an unfavorable outcome with or without bacteriological confirmation, ie, on bacteriological, radiographic or clinical grounds.
Time Frame: From Day 1 to Month 12.
Population: The PP population consisted of the MITT population, excluding patients who were lost to follow-up/withdrawn, had modified/extended treatment for reasons other than unfavourable therapeutic response, did not receive adequate amount of allocated study regimen and patients with major protocol deviations, unless already classified as unfavourable.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 2 Months HRZE / 4 Months HR | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide
Number analyzed (Participants) | 52 | 57 | 47 | 53 | 10
Participants
  Favorable | 38 | 46 | 43 | 52 | 10
  Unfavorable | 14 | 11 | 4 | 1 | 0
Statistical Analysis 1: Comparison: DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide vs DS-TB: 2 Months HRZE / 4 Months HR; Test type: Non-Inferiority — Non-inferiority was assessed using the upper bound of the two-sided 95% CI for the difference between the percentage of patients who are classified as having an unfavourable status on the intervention (6 months moxifloxacin + 200 mg PA-824 + pyrazinamide) and the control regimen (2 months HRZE/ 4 months HR). The intervention was considered to be non-inferior to the control arm if the upper bound 95% CI was < 12%; Treatment difference: unfavourable rate = 6.62, 95% CI 2-sided [-2.15 to 15.40] — (DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide) - (DS-TB: 2 Months HRZE/ 4 Months HR)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Day 1 up to and including 14 days after the last administration of trial medication (up to a maximum of 28 weeks).
Description: The Safety analysis population included all patients in the randomized/assigned to trial medication population set who received at least 1 dose of trial medication. Patients were classified according to treatment received.
Groups:
- DS-TB: 2 Months HRZE/ 4 Months HR: Patients with DS-TB were randomized to receive 150 mg rifampicin + 75 mg isoniazid + 400 mg pyrazinamide + 275 mg ethambutol combination tablets (HRZE) orally once daily from Weeks 1 to 8 during the treatment period. Patients then received 150 mg rifiampicin + 75 mg isoniazid combination tablets (HR) orally once daily from Weeks 9 to 26 during the treatment period. The daily dose of HRZE and HR was calculated based on patients' weight. Patients then entered a follow-up period up to Month 24.
Arm/Group | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide | DS-TB: 2 Months HRZE/ 4 Months HR | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide
All-Cause Mortality (participants affected / at risk) | 4/65 | 3/71 | 3/67 | 2/68 | 1/13
Serious Adverse Events (participants affected / at risk) | 3/65 | 8/71 | 8/67 | 3/68 | 3/13
Other Adverse Events (participants affected / at risk) | 61/65 | 62/71 | 63/67 | 62/68 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide (N=65) | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=71) | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=67) | DS-TB: 2 Months HRZE/ 4 Months HR (N=68) | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=13)
Alanine aminotransferase increased (Investigations) | 0 | 1 | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 3 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lymph node Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Bladder mass (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-TB: 4 Months Moxifloxacin + PA-824 (100 mg) + Pyrazinamide (N=65) | DS-TB: 4 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=71) | DS-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=67) | DS-TB: 2 Months HRZE/ 4 Months HR (N=68) | MDR-TB: 6 Months Moxifloxacin + PA-824 (200 mg) + Pyrazinamide (N=13)
Aspartate aminotransferase increased (Investigations) | 15 | 10 | 15 | 17 | 1
Alanine aminotransferase increased (Investigations) | 13 | 10 | 14 | 11 | 1
Blood uric acid increased (Investigations) | 15 | 11 | 12 | 8 | 1
Gamma-glutamyltransferase increased (Investigations) | 8 | 11 | 11 | 12 | 0
Blood glucose increased (Investigations) | 5 | 2 | 2 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 3 | 3 | 0
Protein urine present (Investigations) | 2 | 1 | 2 | 2 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 11 | 11 | 3 | 2
Vomiting (Gastrointestinal disorders) | 13 | 8 | 6 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 14 | 7 | 5 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 5 | 3 | 2
Toothache (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 24 | 19 | 15 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 20 | 21 | 14 | 22 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 5 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 5 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 5 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 8 | 11 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 6 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 5 | 3 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 4 | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 5 | 6 | 7 | 5 | 2
Dizziness (Nervous system disorders) | 3 | 4 | 7 | 4 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 4 | 3
Somnolence (Nervous system disorders) | 4 | 0 | 1 | 2 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 6 | 3 | 3 | 5 | 1
Proteinuria (Renal and urinary disorders) | 6 | 1 | 3 | 4 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 4 | 8 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 5 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Following 3 deaths associated with hepatotoxicity, recruitment was suspended, followed by a partial clinical hold by the United States Food and Drug Association. The hold was removed but the Sponsor permanently stopped recruitment in December 2016.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting for review and removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02342886/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT02342886/SAP_001.pdf